CLINICAL TRIAL: NCT04065737
Title: A Phase II Open-label, Single Arm Study to Evaluate the Efficacy of Sintilimab(IBI 308) to Prevent High-risk Oral Premalignant Lesions Cancerization
Brief Title: Sintilimab to Prevent High-risk Oral Premalignant Lesions Cancerization
Acronym: STOP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019HNRT01
Record Dates: First submitted 2019-08-05; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-07

CONDITIONS: Oral Cavity Cancer; Mouth Neoplasm; Precancerous Conditions
Keywords: high-risk oral pre-malignant lesions; history of invasive oral cancer; sintilimab
MeSH Terms: conditions — Mouth Neoplasms; Precancerous Conditions | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab (Experimental): Injection; dosage form: 10ml: 100mg; frequency: 200mgQ3W; duration: 8cycles (6 months) or randomization to the date of the first documented oral cancer incidence
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab is a type of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells.
  other name: IBI308
  Other Names: IBI308

SUMMARY:
This is a non-randomized, phase II, open-label study. The goal of this clinical research study is to investigate how well sintilimab works in preventing high-risk oral premalignant lesions cancerization.

DETAILED DESCRIPTION:
this study is a non-randomized, phase II, open-label study. Phase II clinical trials test the safety and effectiveness of an investigational drug or combination of drugs to learn whether it works in preventing or treating a disease.

the purpose of this study is to evaluate the effectiveness of sintilimab in preventing the onset of oral cancer in patients with high-risk oral premalignant lesions, who had oral cancer at least once before.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Histological evidence of oral premalignant lesions (such as leukoplakia and/or erythroplakia). A history of invasive oral cancer or oral cancer in situ, which was histologically confirmed.
3. With at least on high-risk profiles: a. have LOH at 3p14 and/or 9p21; b. pathologically diagnosis with severe dysplasia; c. size of lesions >200mm².
4. Eastern Cooperative Oncology Group Performance Status (ECOG) performance scale: 0-1.
5. Adequate organ and bone marrow function:

   * CBC: absolute neutrophil count (ANC) ≥ 1.5 × 10^9 / L; platelet count (PLT) ≥ 100 × 10^9 / L; hemoglobin content (HGB) ≥ 9.0 g / dL.
   * Liver function: serum total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN.
   * Renal function: serum creatinine (Cr) ≤ 1.5 × ULN.
6. Female subject of childbearing potential should have a negative urine or serum pregnancy test < 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of study therapy through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses > 1 year.
8. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of the study therapy.
9. Voluntarily signed written informed consent form, willing and able to comply with scheduled visits and other requirements of the study.

Exclusion Criteria:

1. Should receive subsequent adjuvant therapy (such as radiotherapy, chemotherapy, immunotherapy)
2. Received major surgery (such as craniotomy, thoracotomy or laparotomy) within 4 weeks of the first dose of study drugs or open wound, ulcer or fracture.
3. Received any anti-tumor therapy (chemotherapy, targeted therapy, tumor immunotherapy or arterial embolization) or radiotherapy within 4 weeks of the first dose of study treatment.
4. Prior therapy with anti-PD-1,anti-PD-L1,anti-CTLA4 antibody.
5. Currently participating in interventional clinical research treatment, or receiving other research medications within 4 weeks prior to the first dose or used research equipment
6. Received any investigational agent within 4 weeks of the first dose of study treatment.
7. Received radiotherapy within 4 weeks of the first dose of study treatment. Received systemic treatment with high-dose corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive drugs within 4 weeks of first dose. Inhaled or topical steroids and adrenal replacement steroid are permitted in the absence of active autoimmune disease.
8. Received attenuated live vaccine within 4 weeks of the first dose of study medication or plan to receive live vaccine during the study period.
9. Subjects with active, known or suspected autoimmune disease such as interstitial pneumonia, uveitis, Crohn's disease, autoimmune thyroiditis. Subjects with cured childhood asthma, type I diabetes mellitus and hypothyroidism only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment.
10. Known history of allogeneic organ or allogeneic hemopoietic stem cell transplantation
11. Known allergic or hypersensitive to docetaxel, any monoclonal antibody or any other components used in their preparation.
12. Uncontrolled concomitant disease, including but not limited to :

    * Active or poorly controlled severe infection
    * Human Immunodeficiency Virus (HIV) infection (HIV antibody positive)
    * Known acute or chronic active hepatitis B (HBV DNA positive) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection
    * Active tuberculosis
    * Symptomatic congestive heart failure (New York Heart Association grade III-IV) or symptomatic, poorly controlled arrhythmia
    * Uncontrolled hypertension (SBP ≥ 160mmHg or DBP ≥ 100mmHg)
    * Prior arterial thromboembolism event, including myocardial infarction, unstable angina, stroke, and transient ischemic attack, within 6 months of enrollment
13. Known history of, or any evidence of active, non-infectious pneumonitis.
14. Other primary malignancy, with the exception of the skin or squamous cell carcinoma of the skin or in situ cervical cancer.
15. Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
oral cancer incidence rate | 2 years
  The proportion of patients who has been diagnosed with oral cavity cancer

SECONDARY OUTCOMES:
clinical response rate of oral premalignant lesions | 2 years
  The proportion of patients whose oral premalignant lesions experienced a Complete Response or a Partial Response
pathologically response rate of oral premalignant lesions | 2 years
  The proportion of patients whose oral premalignant lesions experienced a locally complete response or decrease of histopathological grade
Duration of Response (DoR) of oral premalignant lesions | 2 years
  the time from the date for first documented response of complete response (CR) or partial response (PR) until the date for the first documented response of progressive disease (PD), incidence of oral cancer or death in the absence of progression.
2 year oral-cancer-free survival | 2 years
  time from randomization to the development of histologically confirmed oral cancer or death of any cause, whichever occurs first
Treatment-related Adverse Events (AEs) | From the date of randomization to 90 days after last dose of study treatment
  The grade of AEs and the number of patients with AEs are assessed by the investigator based on CTCAE v4.0 from the date of randomization to 90 days after last dose of study treatment
Overall survival (OS) | 2 year
  OS (per RECIST 1.1 as assessed by the investigator) is defined as the time from the date of randomisation until death due to any cause.
quality of life(QOL) | 2 years
  EORTC QLQ-C30 questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No